CLINICAL TRIAL: NCT05368675
Title: A Pilot Implementation Project of Methadone and Suboxone® for Injecting Drug Users in Ho Chi Minh City, Vietnam
Brief Title: Medication-assisted Treatment for Injecting Drug Users in Vietnam
Acronym: OIT-HCMC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Drug Abuse (U.S. Federal Agency); Expertise France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R01DA033671 (NIH)
Record Dates: First submitted 2022-04-26; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Opioid Use Disorder; HIV Infections
Keywords: medication for opioid use disorder; HIV care
MeSH Terms: conditions — Opioid-Related Disorders; HIV Infections | interventions — Dosage Forms; Methadone; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: medication for opioid use disorder — This is an open-label study. The project proposes to enroll up to 500 opiate dependent individuals entering Medication Assisted Treatment (Methadone or buprenorphine/naloxone) at Go Vap Clinic, HCMC, Vietnam. All participants who appear to meet inclusion criteria and who express interest in drug treatment will be invited to be screened for participation in the research. All participants will receive BDRC sessions (weekly for 12 weeks, monthly thereafter until week 52).
  Other Names: methadone; buprenorphine/naloxone; Behavioral Drug and Risk Counseling

SUMMARY:
HIV continues to spread around the world and new infections in Asia are one of the most important areas for prevention among drug using populations. There is strong and consistent evidence from several countries that while injection drug users (IDU) continue to be a source of new infections, treatment of opiate addiction is an effective prevention measure against further spread. The project evaluated the implementation of a comprehensive opioid use disorder treatment program co-located with an HIV clinic in Ho Chi Minh City, Vietnam. The program includes medication for opioid use disorder (methadone, buprenorphine/naloxone), standardized counseling sessions (BDRC) and HIV testing and care (for people living with HIV).

DETAILED DESCRIPTION:
The drug treatment and HIV research literature of the past 20 years provides strong support for the ability of drug treatment programs to reduce the frequency of drug use, risk behaviors, and incidence of new infections. Findings from these studies also suggest that drug users living with HIV who remain in medication assisted treatment (MAT) and cease drug use are significantly more likely to achieve sustained viral suppression and consequently less likely to transmit HIV. While these data are strong and consistent, they are all derived from countries with highly developed drug and HIV treatment systems. Little data exist regarding the challenges of implementing and integrating new strategies for MAT with linkages to HIV care in resource-limited settings with developing drug and HIV treatment systems.

The proposed project will take place in Ho Chi Minh City (HCMC), Vietnam. In HCMC, 51.8 % of IDUs are estimated to be HIV positive (HCMC Provincial AIDS Committee (PAC) 2009). Methadone maintenance treatment (MMT) for IDUs started as a pilot program in 2008 in Haiphong and HCMC, two of the highest prevalence provinces for injecting drug use. By December 2009, 784 patients were under MMT and 235 were receiving ARV. 30% of patients under MMT are HIV+ (HCMC PAC, 2009). The National goal is to have 80,000 drug users in methadone treatment by 2015. There are currently no buprenorphine/naloxone treatment programs in Vietnam.

The proposed project evaluate the implementation of an MAT program (both methadone and buprenorphine/naloxone) integrated within an HIV treatment setting. This is the first project to establish and evaluate the implementation a buprenorphine/naloxone (Suboxone) treatment program in Vietnam. Participants were enrolled in the integrated MAT program that included drug and risk counseling, and for those who are living with HIV, HIV treatment. Participant'received care for 12 months and then transitioned to community treatment program. The study assessed barriers to implementation.

Primary measures consisted of facilitators and barriers to implementation and retention in MAT generally and Suboxone treatment specifically. The following specific aims are evaluated:

* Establish a new integrated MAT treatment program within and HIV treatment setting in HCMC;
* Evaluate barriers and facilitators to implementation of integrated MAT/HIV treatment;
* Evaluate patient retention and medication adherence in integrated MAT/HIV Care;
* Estimate the costs and benefits of MAT treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* • 18 or more years of age

  * Meets DSM-5 criteria for opiate use disorder
  * Positive urine drug screen for heroin or other opiates
  * Interested in methadone maintenance or Suboxone® treatment for opiate use disorder
  * Injected heroin within past 30 days by self-report, documented by "tracks" or puncture marks
  * Willingness and ability to give informed consent and otherwise participate
  * Provision of adequate locator information

Exclusion Criteria:

* • Clinically significant cognitive impairment, schizophrenia, paranoid disorder, bipolar disorder

  * Known neurological, cardiovascular, renal, or other medical disorder that is likely to impair or make the patient's participation hazardous
  * Physiologically dependent on alcohol, benzodiazepines, or other sedative type drugs
  * Pending legal charges with likely incarceration within next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2013-12-18 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Retention in treatment program at 12 months | 12 months
  Percentage of participants who stay in treatment for 12 months
Adherence in treatment program at 12 months | 12 months
  Missing doses of treatment during time in the study
Cost of 12-month treatment program | 12 months
  Cost of 12 months of the treatment program evaluated with the Drug Abuse Treatment Cost Analysis Program (DATCAP)

SECONDARY OUTCOMES:
Change in substance use from baseline to 12-month follow-up | 12 months
  Evaluation of the change in substance use between baseline and 12-month follow-up assessed by weekly self-report and urine drug screen
Viral load suppression for people living with HIV | 12 months
  Percentage of participants living with HIV with a suppressed viral load at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles P O'Brien, MD, PhD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-05-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT05368675/Prot_SAP_000.pdf
  • Informed Consent Form (2015-11-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT05368675/ICF_001.pdf